CLINICAL TRIAL: NCT00004263
Title: Phase I Study of UCN-01 and Cytarabine (ARA-C) in Patients With Acute Myelogenous Leukemia, and Myelodysplastic Syndromes
Brief Title: Cytarabine and UCN-01 in Treating Patients With Refractory or Relapsed Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM99-165; U01CA062461 (NIH); P30CA016672 (NIH); MDA-DM-99165 (Other: NCI PDQ/UT MD Anderson Cancer Center); NCI-T99-0100; CDR0000067522 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-01-28; First posted 2004-07-26 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; previously treated myelodysplastic syndromes; childhood myelodysplastic syndromes; Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; cytarabine; 7-hydroxystaurosporine; UCN-01
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — 7-hydroxystaurosporine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cytarabine + UCN-01 (Experimental)
  Interventions: Drug: 7-hydroxystaurosporine (UCN-01); Drug: Cytarabine (Ara-C)

INTERVENTIONS:
Drug: 7-hydroxystaurosporine (UCN-01) — 20 mg/m2 IV over 24 hours on days 2-4 of course 1 and over 36 hours beginning on day 2 of subsequent courses. Treatment repeats every 4 weeks for a maximum of 4 courses.
Drug: Cytarabine (Ara-C) — Starting dose 1 g/m2 IV over 24 hours on days 1-4 of each course. Treatment repeats every 4 weeks for a maximum of 4 courses.
  Other Names: ARA-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. UCN-01 may make cancer cells more sensitive to cytarabine.

PURPOSE: Phase I trial to study the effectiveness of cytarabine and UCN-01 in treating patients who have refractory or relapsed acute myelogenous leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of cytarabine when combined with UCN-01 in patients with refractory or relapsed acute myelogenous leukemia or myelodysplastic syndrome. II. Determine the dose limiting toxicity, pharmacokinetics, and pharmacodynamics of this regimen in these patients. III. Assess the antileukemia effect of this regimen in this patient population.

OUTLINE: This is a dose escalation, multicenter study of cytarabine. Patients receive cytarabine IV over 24 hours on days 1-4 of each course. Patients receive UCN-01 IV over 24 hours on days 2-4 of course 1 and over 36 hours beginning on day 2 of subsequent courses. Treatment repeats every 4 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Patients with refractory or relapsed acute myelogenous leukemia, or myelodysplastic syndromes (RAEB or RAEB-T).
2. 2. Performance status of =< 2
3. 3. Signed informed consent indicating that patients are aware of the investigational nature of this study in keeping with the policies of the hospital. The only acceptable consent form is the one attached at the end of this protocol for each participating institution.
4. 4. Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease.
5. 5. Bilirubin and creatinine (or creatinine clearance) should be within institutional normal limits.
6. 6. Patients must have relapsed or failed to respond after high-dose ara-C-based (>=1g/m2/day x 3 days) chemotherapy.
7. 7. Corrected DLCO >50%.
8. 8. Patients with >=3 cardiac risk factors (smoking, hypertension, family history of coronary artery disease, diabetes mellitus, hypercholesterolemia) should have a nuclear medicine stress test.

Exclusion Criteria:

1. 1. The anti-proliferative activity of the experimental drug may be harmful to the developing fetus or nursing infant. Therefore, pregnant and nursing females will be excluded. Patients of childbearing potential should practice effective methods of contraception.
2. 2. Patients who are eligible for allogeneic marrow transplant and who have a donor will be offered transplant.
3. 3. Patients with existing pulmonary diseases, history of coronary artery disease or who have received radiotherapy to the mediastinum.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1999-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Cytarabine + UCN-01 | 4 week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org